CLINICAL TRIAL: NCT06999785
Title: Assessment of the Impact of Increased Production of Reactive Oxygen Species Produced During Repeated Sessions of Hyperbaric Oxygen Therapy in Patients Undergoing Radiotherapy for Neoplasia, on the Occurrence of DNA Damage
Acronym: OXYBAR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 49RC24_0248; 2025-A00812-47 (Other: ANSM)
Record Dates: First submitted 2025-05-05; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Hyperbaric Oxygen; Genotoxicity; Malignancy
MeSH Terms: conditions — Neoplasms | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiation-induced complications (Experimental): The interventions which are specific to the study is a blood test before and after the first oxygen therapy session, as well as after the last session
  Interventions: Biological: Blood test

INTERVENTIONS:
Biological: Blood test — a blood test before and after the first oxygen therapy session, as well as after the last session

SUMMARY:
Hyperbaric Oxygen Therapy (HBOT) is a treatment involving the administration of oxygen at pressures higher than atmospheric pressure, with numerous potential indications such as radiation-induced tissue damage, chronic wounds, and more. HBOT significantly increases the amount of dissolved oxygen in tissues, thereby promoting wound healing.

However, this "hyperoxygenation" may also exert toxic effects, particularly through the production of reactive oxygen species (ROS), which can induce DNA damage and potentially promote mutagenesis, thereby increasing long-term neoplastic risk.

A single HBOT session is associated with a significant increase in ROS production, which may persist for up to 48 hours post-exposure, and is also linked to DNA damage. DNA repair is typically a rapid process, with the activation of protective mechanisms.

The effects of repeated HBOT sessions remain a matter of debate. Reported outcomes range from attenuation of genotoxicity, to exacerbation of DNA damage, or no effect at all (8). In patients with cancer or comorbidities associated with impaired DNA repair capacity, repeated HBOT could be more detrimental, potentially increasing genotoxic effects and cancer risk. This increased oxygen susceptibility in cancer patients has already been observed in normobaric conditions during abdominal surgery, where hyperoxygenation strategies were associated with increased mortality in this subgroup.

A potential pro-carcinogenic effect of HBOT in cancer patients has also been suggested in some case series, though not confirmed by larger studies.

Current literature on HBOT safety remains generally reassuring; however, the possibility of DNA damage and its potential long-term genotoxic consequences cannot be entirely excluded. This question is of particular importance given that many primary indications for HBOT involve patients with a history of malignancy or active cancer

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old)
* Having signed an informed consent form
* Affiliated with or beneficiary of a national health insurance system
* Admitted to the hyperbaric medicine department for HBOT treatment
* Either for a complication related to prior radiotherapy (administered for an underlying neoplastic disease), such as:

Radiation cystitis Radiation proctitis / enteritis Radiation dermatitis Mandibular osteoradionecrosis Or for another indication, without any underlying neoplastic disease

Exclusion Criteria:

* Patients with a contraindication to hyperbaric oxygen therapy (HBOT)
* Pregnant, breastfeeding, or postpartum women
* Patients deprived of liberty by judicial or administrative decision
* Patients undergoing involuntary psychiatric treatment
* Patients under legal guardianship or protective custody

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-11-15 (Estimated)

PRIMARY OUTCOMES:
Correlation between hyperbaric oxygen therapy and DNA damages | Baseline (inclusion, before the first oxygen therapy session), during treatment(just after the first oxygen therapy session) and immediately after treatment (just after the last oxygen therapy session)
  Tail DNA Percentage by the Comet Assay (cellular biology technique, single-cell gel electrophoresis)

SECONDARY OUTCOMES:
reactive oxygen derivatives formation | Baseline (inclusion, before the first oxygen therapy session), during treatment(just after the first oxygen therapy session) and immediately after treatment (just after the last oxygen therapy session)
  8-hydroxy-2'-deoxyguanosine (8-OHdG) plasma levels
reactive oxygen derivatives formation | Baseline (inclusion, before the first oxygen therapy session), during treatment(just after the first oxygen therapy session) and immediately after treatment (just after the last oxygen therapy session)
  isoprostanes (8-isoprostane) plasma levels
Correlation between DNA damage and post-radic wound healing | Baseline (inclusion, before the first oxygen therapy session), during treatment(just after the first oxygen therapy session) and immediately after treatment (just after the last oxygen therapy session)
  Grade difference on the LENT-SOMA scale (Late Effects of Normal Tissues-Subjective, Objective, Management, Analytic)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No